CLINICAL TRIAL: NCT06714370
Title: Real-World Evidence of Effectiveness and Safety of Tirabrutinib in Patients with Relapsed or Refractory Primary Central Nervous System Lymphoma in Taiwan: a Nationwide Study
Acronym: REVEAL
Status: Not yet recruiting | Type: Observational
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: R1128-TIR-04
Record Dates: First submitted 2024-11-05; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Primary Central Nervous System Lymphoma (PCNSL)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to describe the real-world effectiveness and safety of tirabrutinib among relapsed or refractory PCNSL patients in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 18 years of age.
2. r/r PCNSL patient, who has newly started NHI public reimbursement tirabrutinib from 01 June 2024 to 30 June 2025.
3. Have provided voluntary written consent, directly from the subject, or through his/her legal representative for a patient who has died or lacks the capacity to give informed consent

Note: The NHI reimbursement criteria are listed below for reference purposes only. Subject enrollment depends on whether reimbursement has been received.

1. Histopathologically confirmed large B-cell PCNSL.
2. Patients with relapsed or refractory PCNSL previously treated at least 2 cycles of HD-MTX.
3. Exclude HIV infection
4. Exclude Burkitt lymphoma
5. Exclude patients using chemotherapy or monoclonal antibodies at the initiation of tirabrutinib treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient received Taiwan NHI reimbursement
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | At least 9 months for each subject
  objective response rate is defined as the proportion of subjects who respond either Complete response (CR), Partial response (PR), or unconfirmed Complete response (CRu) to therapy, according to International PCNSL Collaborative Group (IPCG) criteria.

SECONDARY OUTCOMES:
Duration of response (DOR) | At least 9 months for each subject
  Duration of response is defined as the time from onset of response* to disease progression or death, wichever occurs earlier.
  *for patients who achieve complete response (CR), partial response (PR), or unconfirmed complete response (CRu), according to IPCG criteria.
Time-to-treatment response (TTR) | At least 9 months for each subject
  Time-to-treatment response was defined as time from newly started tirabrutinib treatment to the first objective tumor response observed for patients who achieved a complete response (CR), partial response (PR), or unconfirmed complete response (CRu), according to IPCG criteria.
Adverse events of special interest (AESIs) | At least 9 months for each subject
  Drug-related adverse events for treatment interruption, dose reduction, and discontinuation of tirabrutinib: febrile neutropenia (grade≥3), thrombocytopenia with hemorrhage (grade 3), neutropenia (grade 4), thrombocytopenia (grade 4), interstitial lung disease (grade≥2), skin disorder (grade≥2), hematotoxicity (grade≥3, other than events described above) and nonhematological toxicity (other than interstitial lung disease and skin disorder, grade≥3) (the grading will be according to CTCAE v5.0.) important identified risks: infection, severe skin disorder, bone marrow depression, hypersensitivity, interstitial lung disease (ILD), hepatic dysfunction, hemorrhage, arrhythmia.
Clinical laboratory test | At least 9 months for each subject
  Clinical laboratory tests (hematology, blood biochemistry, urinalysis, etc.) will be summarized with dexcriptive statistics. The change from baseline will be presented also, if possible.
Treatment-emergent adverse events (TEAEs) | At least 9 months for each subject
  in this study, an AE is defined as any unfavorable or unintended injury/disease or sign (including an abnormal laboratory finding) in a subject administered tirabrutinib, regardless of causality. AE also includes suspected transmission of infectious agents by tirabrutinib. TEAE is defined as an AE that began after the start of tirabrutinib treatment. Concurrent disease at the start of tirabrutinib treatment that has worsened during tirabrutinib treatment for the subject is also included. worsening of the primary disease is not an TEAE. all severity of AEs will be graded according to CTCAE v5.0. All AE that are not considered serious AE are not-serious AE.
Overall survival (OS) | At least 9 months for each subject
  overall survival is defined as time from newly started tirabrutinib treatment to death.
Progression-free survival (PFS) | At least 9 months for each subject
  Progression-free survival is defined as time from newly started tirabrutinib treatment to either first evidence of progression disease (PD), according to IPCG criteria, or death.

OTHER OUTCOMES:
ECOG Performance Status Scale | At least 9 months for each subject
  the ECOG performance status scale was developed by the Eastern Cooperative Oncology Group, now the ECOG-ACRIN Cancer Research Group, and published in 1982. From Grade 0 fully active, able to carry on all pre-disease performance without restriction, to Grade 5 Dead. ECOG performance status scale will be listed and summarized by number and percentage by scoring categories.
Clinical usage and pattern of tirabrutinib | At least 9 months for each subject
  For the clinical usage and pattern of tirabrutinib, exposure duration and daily dose for tirabrutinib during study period will be listed for each subject and summarized with descriptive statistics.
Ratio of the premedications for infection and skin-related disorders | At least 9 months for each subject
  the premedications for infection and skin-related disorders will be listed and tabulated with number and percentage.

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol